CLINICAL TRIAL: NCT03927391
Title: Effect of a Reduced Dose on Cognitive Side Effects of Enzalutamide in Frail (Metastatic) Castration-resistant Prostate Cancer Patients (REDOSE)
Brief Title: Effect of a Reduced Dose Enzalutamide in Frail (m)CRPC Patients on Cognitive Side Effects
Acronym: REDOSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REDOSE
Record Dates: First submitted 2019-03-29; First posted 2019-04-25 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: enzalutamide; cognitive side effects
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — enzalutamide

STUDY DESIGN:
Intervention Model Description: Normal enzalutamide dose versus reduced dose in two patient groups
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor does not know the treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reference (normal) dose (Active Comparator): Normal dose of enzalutamide (160mg once daily)
  Interventions: Drug: Enzalutamide
- test (reduced) dose (Experimental): Reduced dose of enzalutamide (120mg once daily)
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — enzalutamide treatment

SUMMARY:
Prostate cancer is the most commonly diagnosed cancer among men in Western countries. When the disease recurs as castration-resistant prostate cancer (CRPC) it is associated with a median overall survival of approximately 2 years with significant decrement in quality of life due to additional cancer-specific and treatment-induced morbidity. Palliative agents currently used in the CRPC setting include the 2nd generation hormonal agents abiraterone acetate and enzalutamide but also radium-223, docetaxel and cabazitaxel. Choices for treatment strategies are based on multiple factors such as age, co-morbidity and drug toxicity profile. The side effect profile of enzalutamide is associated with central nervous system (CNS side effects) such as fatigue and depression. The mechanism for these side effects is not yet fully understood, but it was shown in rodent studies that enzalutamide and its active metabolite penetrate into the CNS. This might cause the CNS side effects that were later seen in the phase 1 study where fatigue was found to be a dose-dependent adverse event. After dose reductions the symptoms resolved. This was also found in a retrospective study of Japanese metastatic CRPC (mCRPC) patients (n=345) in which the side effects malaise and nausea decreased remarkably after dose reduction. However, no exposure-response relation was observed in the study of Gibbons et al. Additionally, based on the data of the phase 1 trial of enzalutamide it can be suggested that a minimum trough concentration of 5.0 mg/L could be considered as a target for exposure to enzalutamide. In particular, frail (m)CRPC patients are more prone to develop CNS side effects on enzalutamide. The investigator's hypothesis is that dose reduction to 75% (120mg) can be safely done to treat (m)CRPC in these patients with preserving optimal efficacy and less CNS side effects.

ELIGIBILITY:
Inclusion Criteria:

* Frailᵃ male patients with prostate cancer who will start treatment with enzalutamide within label
* Age at least 18 years
* Patient who are able and willing to give written informed consent prior to screening
* Patients from whom it is possible to collect blood samples
* Patients who are willing to answer the questionnaires and test
* Life expectancy of > 6 months
* Capable of understanding and answering Dutch tests and questionnaires, as determined by the investigator

ᵃ Frail is defined as:

* a score on the comprehensive G8 assessment with cut-off ≤14 points and
* score ≥grade 1 for Central Nervous Disorders according to the Common Toxicity Criteria Adverse Event (CTCAE) criteria, of one of the following: Fatigue, Concentration impairment, cognitive disturbance, amnesia, depressed level of consciousness, memory impairment, hypersomnia.

Exclusion Criteria:

* change in dose of opioids/sedatives/benzodiazepines during last 2 weeks before study)
* Use of psychostimulants such as methylphenidate within 1 week of start of study
* Diagnosed with medical conditions that affect cognition: Dementia, Alzheimer disease, Parkinson's disease, psychiatric disorders that affect cognition other than depression or anxiety complaints related to the disease
* Active infection or other comorbidities that may contribute to REDOSE, February 2019 Page 7 of 53 fatigue or cognition change within 4 weeks of study entry
* Clinical relevant anaemia
* MoCa score <20
* Hypersensitivity to the active substance or to any of the excipients.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer is only prevalent in the male population
Enrollment: 57 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
To determine the change in the CNS side effect fatigue* in frail (m)CRPC patients treated with a reduced dose of enzalutamide (120mg OD) compared to the standard dose of enzalutamide (160mg OD) after 6 weeks of treatment. | 6 weeks
  *fatigue is measured by the self-reported FACIT-fatigue questionnaire version 4 (Dutch version). Functional Assessment of Chronic Illness Therapy-Fatigue. 13-items are scored on a 5-point scale. All items except items 7 (I have energy) and 8 (I am able to do my usual activities) are reverse-scored before item scores are summed to obtain a total score (range 0-52). Higher scores reflect less fatigue.4 (Dutch version): Functional Assessment of Chronic Illness Therapy-Fatigue. 13-items are scored with a total score ranging 0-52. Higher scores reflect less fatigue.

SECONDARY OUTCOMES:
To determine the decrease in the CNS side effect fatigue in frail (m)CRPC patients treated with a reduced dose of enzalutamide (120mg OD) compared to the standard dose of enzalutamide (160mg OD) after 12 weeks, and 24 weeks of treatment. | 12 weeks and 24 weeks
  fatigue is measured by the self-reported FACIT-fatigue questionnaire version 4 (Dutch version). Functional Assessment of Chronic Illness Therapy-Fatigue. 13-items are scored on a 5-point scale. All items except items 7 (I have energy) and 8 (I am able to do my usual activities) are reverse-scored before item scores are summed to obtain a total score (range 0-52). Higher scores reflect less fatigue.
To determine the impact of cognition impairment in quality of life in frail (m)CRPC patients treated with a reduced dose of enzalutamide (120mg OD) compared to the standard dose of enzalutamide (160mg OD). | 6, 12 and 24 weeks
  The impact of cognition impairment in quality of life is measured by the self-repored FACT-cog questionnaire. FACT-cog: Functional Assessment of Cancer Therapy - For patients with Cognitive function issues. There are 4 subscale scores (perceived cognitive impairments (range 0-72), impact of perceived cognitive impairments on quality of life (range 0-16), comments from others (range 0-16) and percieved cognitive abilities (range 0-28). All subscale scores are summed to derive a total score. The higher the score, the better quality of life.
To determine cognition impairment in frail (m)CRPC patients treated with a reduced dose of enzalutamide (120mg OD) compared to the standard dose of enzalutamide (160mg OD). | 6, 12 and 24 weeks
  cognition impairment is measured by the MoCA test. Montreal Cognitive Assessment, is a test for cognition. It covers 8 tasks: attention and concentration, executive functions, memory, language, visuospatial abilities, abstract thinking, calculating abilities and orientation. The maximum score is 30 points. The higher the score, the better the cognition is.
To evaluate changes in depression score in frail (m)CRPC patients treated with a reduced dose of enzalutamide (120mg OD) compared to the standard dose of enzalutamide (160mg OD). | 6, 12 and 24 weeks
  Geriatric depression scale 15 (GDS-15): 15 question using an ordinal score (yes/no). Total score: maximum 15 points. A score of 0 to 5 is normal. A score greater than 5 suggests depression.
To correlate exposure (Ctrough) of enzalutamide and n-desmethylenzalutamide to the CNS side effects. | 6, 12 and 24 weeks
  Correlations of Ctrough and CNS side effects
To determine the percentage (%) of subjects that remained on the allocated dose level until the end of the study. | 6, 12 and 24 weeks
  % subjects that without dose reductions or dose increments
To evaluate the effect of dose reduction on treatment efficacy according to prostate cancer working group 3 (PCWG3). | 6, 12 and 24 weeks
  Effect of dose reduction (120mg) on treatment efficacy

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - CWZ, Nijmegen
  - Radboudumc, Nijmegen
  - Franciscus Gasthuis en Vlietland hospital, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boerrigter E, Overbeek JK, Benoist GE, Somford DM, Hamberg P, Tol J, Scholtes B, Willemsen AECAB, Buffart LM, Kessels RPC, Mehra N, van Oort IM, van Erp NP. A Prospective Randomised Trial to Determine the Effect of a Reduced Versus Standard Dose of Enzalutamide on Side Effects in Frail Patients with Prostate Cancer. Eur Urol Oncol. 2024 Dec;7(6):1376-1383. doi: 10.1016/j.euo.2024.02.009. Epub 2024 Mar 13. PMID 38485614